CLINICAL TRIAL: NCT04275050
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB3303 Tablets
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB3303 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3303-I-0001
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-06

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3303 Tablet (Experimental): TQB3303 Tablet administered orally once. Then TQB3303 Tablet administered orally, once daily in 28-day cycle after 7 days of first administration.
  Interventions: Drug: TQB3303

INTERVENTIONS:
Drug: TQB3303 — TQB3303 tablet is a small molecule oral drug inhibiting cyclin-dependent kinases 4 and 6 (CDK4 / 6).

SUMMARY:
TQB3303 tablet is a small molecule oral drug inhibiting cyclin-dependent kinases 4 and 6 (CDK4 / 6). Based on current research, overexpression of positive regulatory proteins in the cell cycle is one of the important reasons for resistance to endocrine therapy. CDK4 / 6 is the key regulators of the cell cycle inhibiting tumor cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* 1.≥ 18 years old. 2. Histologically or cytologically confirmed advanced malignant solid tumors, without conventional treatment methods or fail or relapse after treatment.

  3.Has at least one measurable lesion (based on RECIST 1.1) or bone metastases. 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥12 weeks.

  5. Adequate organ system function. 6.Understood and signed an informed consent form. 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

* 1. Has diagnosed and/or treated additional malignancy with the exception of cured basal cell carcinoma of the skin and cervical carcinoma in situ.

  2. Has received cytotoxic chemotherapy in 4 weeks, or mitomycin C or nitrosourea in 6 weeks.

  3. Has received any anti-tumor treatment such as hormone therapy, radioimmunotherapy, molecular targeted therapy, immunotherapy or other biological therapy within 4 weeks.

  4. Has received other CDK4 / 6 inhibitors. 5. Has known spinal cord compression, cancerous meningitis, newly diagnosed central nervous system metastasis or brain metastases with stable symptoms less than 4 weeks; asymptomatic and stable imaging without corticosteroid treatment.

  6.Has received stem cell or bone marrow transplant. 7.Has multiple factors affecting oral medication. 8.Has uncured wounds or fracture, except of pathological fracture with bone metastases patients.

  9.Has uncontrolled cardiovascular disease. 10.Has received CYP3A4 inhibitors or inducers during the screening period and during the trial.

  11.Has drug abuse history that unable to abstain from or mental disorders. 12.urinary protein ≥ ++, and the 24-hour urine protein quantification > 1.0 g. 13. Has active hepatitis B or C. 14. Has a history of autoimmune disease, immunodeficiency. 15. Hypersensitivity to TQB3303 or its excipient. 16. Has participated in other clinical trials within 4 weeks before participating in this trial.

  17. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the following toxic reaction relate to the drug after treatment within 28 days ：III °or above of non-hematological toxicity, IV° hematological toxicity , III ° neutropenia associated with fever, III ° thrombocytopenia with bleeding， III ° QTc interval extended

SECONDARY OUTCOMES:
Cmax | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on single dose; Hour 0 of day 7,day 14,day21 on multiple dose and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on multiple dose of day 28.
  Cmax is the maximum plasma concentration of TQB3303 or metabolite(s).
Tmax | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on single dose; Hour 0 of day 7,day 14,day21 on multiple dose and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3303 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on single dose; Hour 0 of day 7, day 14, day21 on multiple dose and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3303 by assessment of area under the plasma concentration time curve from zero to infinity.
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciencesand Peking Union Medical College, Beijing, Beijing Municipality, China